CLINICAL TRIAL: NCT02500420
Title: Study of Hypertrophic Cardiomyopathy Under Stress Conditions. Concordance Between Two Complementary Tests: Stress MRI and Exercice Stress Echocardiography
Acronym: CMHStress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9517
Record Dates: First submitted 2015-03-23; First posted 2015-07-16 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; Stress MRI; Cardiac MRI; Stress echocardiography; T1 mapping; 2D strain
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis examens (Other): * Cardiac MRI: is usually recommended in the diagnosis or in the follow-up of the disease. The MRI will respect the standard protocol: cineMRI sequences, perfusion sequences, LGE sequences at 10 minutes after gadolinium injection. The investigators will realize some additional sequences: T1 mapping before and after gadolinium injection to study the diffuse fibrosis and stress perfusion sequences after injection of a vasodilatator (Persantine°).
  * Exercice stress echocardiography: is realized almost systematically in all the diagnosis of HCM and it's very informative. The investigators will research left ventricular dysfunction: in particular segmentary hypokinesia and anomalies of deformation parameters (2D Strain) and the development of a dynamic left ventricular outflow obstruction or a mitral regurgitation at exercice.
  Interventions: Other: Diagnosis examens

INTERVENTIONS:
Other: Diagnosis examens — * Cardiac MRI: is usually recommended in the diagnosis or in the follow-up of the disease. The MRI will respect the standard protocol: cineMRI sequences, perfusion sequences, LGE sequences at 10 minutes after gadolinium injection. The investigators will realize some additional sequences: T1 mapping before and after gadolinium injection to study the diffuse fibrosis and stress perfusion sequences after injection of a vasodilatator (Persantine°).
  * Exercice stress echocardiography: is realized almost systematically in all the diagnosis of HCM and it's very informative. The investigators will research left ventricular dysfunction: in particular segmentary hypokinesia and anomalies of deformation parameters (2D Strain) and the development of a dynamic left ventricular outflow obstruction or a mitral regurgitation at exercice.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a primitive myocardic disease and the first of genetic cardiac diseases. The definition of HCM is an increase of the myocardial thickness of the left ventricle (LV) wall without any other causes of hypertrophy. It's characterized by an important heterogeneity of prognosis and clinical expression going from a asymptomatic state until the devastating sudden death occurring in a young person.The diagnosis of HCM is definite by a myocardial thickness greater or equal to 15mm (or 13mm if there is a familial history).This hypertrophy is often accompanied by other abnormalities detected by echocardiography: dynamic left ventricular outflow obstruction at rest or stress, mitral regurgitation …Now, the current challenge is to determine the prognosis factors of the disease that could help to identify the patients with high risk of sudden death. Some prognosis factors are knowed and used in the calculation of a new risk score. This risk score allows to estimate the risk of sudden death at 5 years and propose depending on the result, the implantation of a defibrillator for primary prevention.The physiopathological mechanism of HCM is very complex and still misunderstood. Myocardial fibrosis could be a major mechanism of the disease evolution. Indeed, fibrosis is responsible of scar areas where ventricular tachycardia may develop. Moreover, if the fibrosis is very extensive, it can be the responsible of a systolic or diastolic dysfunction of the left ventricle leading to heart failure.Myocardial ischemia caused by a microvascular dysfunction is now recognized as an important mechanism of the disease evolution. Acute ischemic events could be a trigger of malignant arrhythmia whereas chronic ischemia leads to fibrosis.Left ventricle function is long time preserved in HCM. Segmentary hypokinesia corresponding to extensive fibrosis appears at a very advanced stage of the disease. Exercice stress echocardiography permits to detect myocardial ischemia caused by microvascular dysfunction in the HCM before the fibrosis apparition. Moreover the investigators suggest to study the deformation parameters by speckle tracking or 2D strain witness of a contractile LV dysfunction before the apparition of segmentary hypokinesia.Magnetic resonance imaging (MRI) is now recognized as the more sensible technique to identify focal myocardial fibrosis resulting in areas of late gadolinium enhancement (LGE). LGE is frequent in HCM and his extension is correlated with the severity of the hypertrophy and the risk of sudden death. Myocardial ischemia is detected by hypoperfused defects in the perfusion sequences and as LGE, is correlated with the degree of hypertrophy. Some studies using stress MRI with vasodilatator agent show inductible hypoperfused areas correlated to the degree of hypertrophy. T1 mapping is a new hopeful sequence of MRI permitting to detect the diffuse and early myocardial fibrosis. Some studies show that T1 mapping values are reduced in the areas of LGE in HCM but also in areas without LGE which reflects the presence of new fibrosis.The objective of study is to compare these two imagery techniques in order to detect ischemia and fibrosis. These techniques are usually used in the diagnosis or the monitoring of the disease. The investigators propose to realize an exercise stress echocardiography to study: the segmentary kinetic of the left ventricle and the 2D strain and a stress MRI to study the LGE, the stress perfusion and the T1 mapping.Actually the investigators consider that LGE is a risk factor of the disease (although not yet involved in the calculation of the risk of sudden death) and need to be study in each MRI realized for HCM. From the same way, the investigators suggest to follow patients to determine if the abnormalities detected by these two techniques and particularly 2D strain abnormalities, stress myocardial ischemia and T1 mapping abnormalities are prognosis factors of the disease and appear more precociously than LGE.

ELIGIBILITY:
Inclusion Criteria:

* The patient is adult (> or = 18 years) and informed.
* He's agree for a 24-month follow-up.
* The patient must be member or beneficiary of a health insurance system.
* He must have a clear diagnosis of HCM defined by a left ventricular hypertrophy in tranthoracic echocardiography (superior to 15mm or 13mm if there is a familial history) without other causes of hypertrophy (severe hypertension, aortic stenosis, amyloidosis or fabry disease, ..)

Exclusion Criteria:

* The patient is under safeguarding justice, tutorship or curatorship.
* The patient formalizes his opposition.
* It's impossible to give enlightened information.
* The patient doesn't read French.
* The patient is pregnant or breastfeeding.
* Contraindication to the realization of a MRI (defibrillator, no-MRI compatible PMK, claustrophobia,..)
* Contraindication to the Persantine° injection (asthma, high degree block, ..)
* Contraindication or impossibility to realize a stress echocardiography.
* Comorbidity that can be responsible of the studied anomalies: coronaropathy, myomectomy, multicomplicated diabetes, …

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with myocardial ischemia in MRI without segmental wall-motion abnormality in exercise echocardiography. | Baseline
  In MRI, myocardial ischemia is defined as the presence of an hypoperfused defect in the stress perfusion sequences. Presence of hypoperfused defects: YES / NO; if YES: number of segments affected among the 17-segments bullseye plot of the left ventricle (LV).In echocardiography, segmental wall-motion abnormality is recognized as significant if it affects more than 10% of the left ventricle. Presence of a significant wall-motion abnormality at exercise: YES / NO; if YES: number of LV segments affected.

SECONDARY OUTCOMES:
Number of patient with myocardial ischemia in MRI (same definition as defined in the primary outcome measure) and presence of late gadolinium enhancement (LGE) in MRI. | Baseline
  LGE is defined as the presence of an hyperintense signal in the LGE sequences at 10 minutes in at least one segment among the 17-segments bullseye plot of the LV. Presence of LGE: YES / NO; if YES: extension calculated with the number of affected segments among the 17-segments bullseye plot of the LV .
Number of patient with myocardial ischemia in MRI (same definition as defined in the primary outcome measure) and elevation of T1 mapping before gadolinium injection or decrease of T1 mapping after gadolinium injection. | Baseline
  A significant increase of T1 mapping before gadolinium injection is retained for a rate higher than 1050. A significant decrease of T1 mapping after gadolinium injection is retained for a rate lower than 350.
Number of patient with myocardial ischemia in MRI (same definition as defined in the primary outcome measure) and alteration of global and segmentary longitudinal speckle tracking or "2D Strain" at rest and exercise in echocardiography. | Baseline
  We retain a significant alteration of 2D strain for a rate lower than 16%. The segmental analysis is realized with the 17-segments bullseye plot of the LV.
Time between inclusion and the occurence of an interest event like: hospitalization for cardiovascular reasons or cardiovascular death. | 24 months after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Arnaud de Villeneuve - CHRU de Montpellier, Montpellier, France